CLINICAL TRIAL: NCT05962190
Title: The Effect of Short-term Overconsumption of Specific Dietary Nutrients on Liver and Adipose Tissue Metabolism.
Brief Title: Short-term Fat Overfeeding on the Effects of Liver Metabolism
Acronym: FOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 211172
Record Dates: First submitted 2023-03-20; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-03

CONDITIONS: Liver Fat; Cardiac Function; Lipid Disorder; Adiposity
MeSH Terms: conditions — Fatty Liver; Lipid Metabolism Disorders; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat, high SFA (Experimental): ~60% of total energy is from fat, of which ~45% is from SFA, ~55% is from PUFA
  Interventions: Behavioral: Diet
- High fat, high UFA (Experimental): ~60% of total energy is from fat, of which ~25% is from SFA, ~75% from UFA
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — High fat (~60% of total energy intake) diet enriched with either SFA or UFA

SUMMARY:
Despite work showing the overconsumption of saturated fatty acids (SFA) to be metabolically deleterious, debate continues about whether there is a link between SFA and cardiovascular disease risk. To explore this, we are undertaking a human in vivo parallel-design study, comparing two isocaloric high-fat diets; one enriched with SFA and the other enriched with unsaturated fatty acids (UFAs), to determine the impact of dietary fat composition on postprandial metabolism, liver fat, cardiac fat and cardiac function.

DETAILED DESCRIPTION:
The investigators will recruit men and women with no medical condition or relevant drug therapy that affects lipid, glucose or liver metabolism.

Purpose and design:

The investigators are asking the research question: "How does the amount and type of fat consumed, influence liver fat content, cardiac function and postprandial fatty acid and liver fat metabolism when someone is not gaining or losing body weight?"

To address this research question investigators want to undertake detail physiological studies, in a parallel dietary intervention, where individuals will have an MRI/S scans to assess liver fat, cardiac fat and cardiac function, along with a postprandial study day to assess how their metabolic response to a experimental test meal, before and then 28 days after consumption of a eucaloric, high fat intervention diet that will be either enriched in saturated or unsaturated fat.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged ≥18 or ≤65 years.
* Body Mass Index ≥19 ≤35 kg/m2
* No medical condition or relevant drug therapy that is known to affect liver or adipose tissue metabolism.
* Weight stable for the previous 3 months

Exclusion Criteria:

* The participant is unwilling or unable to give informed consent for participation in the study. - Aged ≤18 or ≥65 years
* Body Mass Index ≤19 or ≥35kg/m2
* Blood haemoglobin <135mg/dL for men and <120mg/dL for women
* Donated (or lost) ≥250 ml of blood in the previous two months.
* On a weight loss diet or have decreased their body weight by >5% in the previous 3 months.
* Have increased their body weight by >5% in the previous 3 months.
* Any metabolic condition or relevant drug therapy
* Current smoker
* History of alcoholism or a greater than recommended alcohol intake (>30 g of alcohol daily for men and >20 g of alcohol daily for women)
* Haemorrhagic disorders
* Anticoagulant treatment
* History of albumin allergy
* Pregnant or nursing mothers
* Women prescribed any contraceptive agent or device including oral contraceptives, hormone replacement therapy (HRT) or who have used these within the last 12 months History of severe claustrophobia
* Presence of metallic implants, pacemakers, or are unwilling to remove any piercings
* History of an eating disorder or any other psychological condition that may affect the participant's ability to adhere to study intervention/experimental diets.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Liver fat | Pre- and after approx 28 days of consuming interventional diet
  Changes in intrahepatic triglyceride, as measured by MRI

SECONDARY OUTCOMES:
Postprandial plasma biochemistry | Pre- and after approx 28 days of consuming interventional diet
  Changes in postprandial plasma triglycerides, glucose, insulin over 6 hours following consumption of a standardized experimental test meal

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Hodson, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No